CLINICAL TRIAL: NCT05914064
Title: Gravitas Feeding Tube System Placement Validation in Neonates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gravitas Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRD-04-1645-01
Record Dates: First submitted 2023-04-18; First posted 2023-06-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nasogastric Tube

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Gravitas FT System (Experimental)
  Interventions: Device: Gravitas FT and Gravitas FT Monitor guidance

INTERVENTIONS:
Device: Gravitas FT and Gravitas FT Monitor guidance — FT placed with guidance from the Gravitas FT system

SUMMARY:
The purpose of this study is to validate the Gravitas Feeding Tube System Placement Algorithm for NICU patients and to evaluate the safety and effectiveness of the Gravitas Feeding Tube in the neonate population for the administration of nutrition, fluids and medications.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the Newborn Intensive Care Unit or on the general medical floor requiring a 5-8 Fr NG tube. The desired size of the feeding tube should be determined clinically, and the Gravitas 5-8 Fr Feeding Tube should only be placed if that size is appropriate.
* Age at enrollment: 0 to 2 years post-partum. Can be up to 15 weeks preterm (gestational age ≥ 25 weeks).
* Suitable to start or continue gastric enteral feeding, or otherwise clinically indicated to receive a feeding tube.
* If enteral nutrition has already been initiated, the orogastric/nasogastric feeding tube may be replaced with a Gravitas Feeding Tube.
* Ability to have a legally authorized representative provide informed consent Both neonates on a ventilator (non-invasive or invasive ventilation) or not requiring a ventilator are eligible for this study.

Exclusion Criteria:

* Known major upper airway malformation (e.g. tracheoesophageal fistula)
* Known major GI malformation (e.g. malrotation, esophageal atresia, etc.)
* History of gastrectomy or esophagectomy
* Expected survival of less than one week
* Neonate on ECMO
* Deemed unsuitable for enrollment in study based on the judgement of the site principal investigator for any other reason
* Requirement for post-pyloric feeds (distal to stomach)
* Infant has a basilar skull fracture

Ages: 0 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of device and procedure-related adverse events that occur while the feeding tube is within a subject. The number and type of adverse events will be collected. | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lucile Packard (Stanford) Children's Hospital, Stanford, California
  - Memorial Health University Medical Center, Savannah, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Women & Infants Hospital, Rhode Island, Providence, Rhode Island
  - University of Virginia Children's Health, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No